CLINICAL TRIAL: NCT06532591
Title: Neoadjuvant or Adjuvant Cadonilimab (PD-1/CTLA-4 Bispecific Antibody) Plus Chemotherapy in Patients With Resectable Stage IB (≥4 cm) to IIIB(N2) PD-L1 Negative Non-small Cell Lung Cancer
Brief Title: Neoadjuvant/Adjuvant Cadonilimab Plus Chemotherapy in Patients With Resectable PD-L1 Negative NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Juan LI, MD, Doctor of Oncology, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK2024001
Record Dates: First submitted 2024-04-10; First posted 2024-08-01 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: NSCLC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Cadonilimab +Paclitaxel/ Albumin-bound paclitaxel +Carboplatin (Experimental): Drug:Cadonilimab +Paclitaxel/ Albumin-bound paclitaxel+Carboplatin neoadjuvant chemotherapy[Cadonilimab, 10mg/kg ,d1,q3w; Paclitaxel 175mg/m2 ivgtt d1/Albumin-bound paclitaxel 260mg/m2,ivgtt(>30min) ,d1,q3w; carboplatin AUC 5 ivgtt d1, q3w] for 3 cycles.The patient was evaluated after 3 cycles of neoadjuvant chemotherapy. The surgery was performed 3-6 weeks after the completion of neoadjuvant chemotherapy. After surgery patients could receive up to 12 months of adjuvant chemotherapy.
  Interventions: Drug: cadonilimab+paclitaxel/albumin-bound paclitaxel+carboplatin

INTERVENTIONS:
Drug: cadonilimab+paclitaxel/albumin-bound paclitaxel+carboplatin — PD-1/CTLA-4 bispecific antibody，Cadonilimab 10mg/kg IV, q3w, paclitaxel 175mg/m2 or albumin-bound paclitaxel 260mg/m2 ivgtt d1, q3w carboplatin AUC 5 ivgtt d1, q3w

SUMMARY:
The purpose of this study is to observe and evaluate the efficacy and safety of cadonilimab combined with chemotherapy in patients with resectable IB (≥ 4cm) - IIIB (N2) stage PD-L1 negative non-small cell lung cancer

DETAILED DESCRIPTION:
This study is design to prospectively investigate the safety and efficacy of cadonilimab combined with chemotherapy in patients with resectable IB (≥ 4cm) - IIIB (N2) stage PD-L1 negative NSCLC. This is a single-institution, single-arm phase 2 clinical trial. Patients will receive 3 cycles of neoadjuvant chemotherapy. The surgery was performed 3-6 weeks after the completion of neoadjuvant chemotherapy. After surgery patients could receive up to 12 months of adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 70 years
* Patients with non-small cell lung cancer diagnosed by pathologic histology or cytology, and the primary focus or lymph node metastasis test is clearly negative for EGFR/ALK/ROS1;
* Tumor tissue PD-L1 expression TPS <1%
* Patients with resectable stage IB (≥4 cm) to IIIB (N2) NSCLC (according to the staging criteria of the American Joint Committee on Cancer, 7th edition)
* Eastern Cooperative Oncology Group performance-status score of 0 or 1
* No previous anticancer therapy
* Patients had to have measurable disease according to the Response Evaluation Criteria in Solid Tumors, version 1.1, and pretreatment tumor tissue available to assess the expression of programmed death ligand 1 (PD-L1)
* Normal function of major organs

Exclusion Criteria:

* Patients with large cell carcinoma and mixed cell lung cancer, mixed with small cell lung cancer components;
* Presence of locally advanced unresectable or metastatic disease;
* Patients in whom imaging shows that the tumor has invaded a vital vascular perimeter or in whom, in the judgment of the investigator, there is a high likelihood that the tumor will invade a vital vessel and cause a fatal hemorrhage during the follow-up study; or patients in whom there is a significant cavitating or necrotic tumor in the lung;
* Has undergone any systemic anticancer therapy for NSCLC, including cytotoxic drug therapy, immunologic drug therapy, experimental therapy;
* Has undergone localized radiotherapy for NSCLC;
* Patients who have had a cancer other than NSCLC in the five years prior to the start of treatment in this study. Patients with cancers other than NSCLC within five years prior to the start of treatment in this study. Excluding cervical carcinoma in situ, cured basal cell carcinoma, and epithelial tumors of the bladder [including Ta and Tis];
* Allergy to cardunculizumab or any component of the chemotherapeutic agent;
* Patients with the presence of any severe and/or uncontrolled disease
* Previous interstitial lung disease, drug-induced interstitial disease, radiation pneumonitis requiring hormonal therapy, or any active interstitial lung disease with clinical evidence;
* Patients who have had a cerebrovascular accident (including temporary ischemic attack) and pulmonary embolism within 6 months;
* Current peripheral neuropathy of ≥ CTCAE grade 2, except as a result of trauma; patients requiring total right lung resection; subjects who have had major surgery or severe trauma and whose effects of surgery or trauma have resolved less than 14 days prior to enrollment
* Patients who are participating in another clinical study or who are less than 4 weeks from the end of treatment in the previous clinical study;
* History of known severe hypersensitivity reactions to other monoclonal antibodies;
* Pregnant or lactating women;
* Previous history of definite neurologic or psychiatric disorders, including epilepsy or dementia;
* Patients who, in the judgment of the investigator, may have other factors that could lead to termination of the study, such as other serious medical conditions or serious laboratory abnormalities or other family or social factors that could affect the safety of the subject or the collection of trial data and samples.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Major pathological response (MPR) | At time of surgery
  MPR is defined as the percentage of residual viable tumour cells (%RVT) in the tumour bed of no more than 10%.

SECONDARY OUTCOMES:
Pathologic complete response (pCR) | At time of surgery
  pCR is defined as no invasive and no in situ residuals in lung and nodes
Objective response rate (ORR) | Up to 1 year
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1
Event free survival at 24 months (EFS24) | Up to 2 year
  EFS24 is defined as patient outcomes were evaluated at diagnosis and in the subsets of patients achieving event-free status at 24 months from diagnosis.
Treatment-Emergent Adverse Event (TEAE) | Up to 2 year
  TEAE is defined as any adverse and unexpected change in body structure, function, or chemistry or any exacerbation of an existing condition (i.e., any clinically significant adverse change in frequency and/or intensity) during treatment. The type, frequency, and severity of TEAE will be assessed during treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial Tumor Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No